CLINICAL TRIAL: NCT03963557
Title: Cognitive Function and Body Mass Index in Children and Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: IREC035
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Obesity, Childhood; Obesity, Adolescent; Cognitive Orientation
MeSH Terms: conditions — Pediatric Obesity; Orientation, Spatial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: BMI 5th percentile to less than the 85th percentile
- Overweight/Obese participants: BMI 85th percentile or more

SUMMARY:
The child will complete computerized tasks and paper-pencil test, and will be presented with symbols, letters, or numbers on a computer screen and asked to respond by pressing a button on the computer. Before each task a researcher will explain the instructions of the task and assess if the child needs a break before completing the next task. While the child is completing computerized tasks, the parent/guardian will be asked to fill out paper-pencil questionnaires about the child and to sign a release of medical information form so that we can study how physical markers of health effect cognition.

ELIGIBILITY:
Inclusion Criteria:

* Local population (based on ethnicity)
* Healthy or overweight/obese

Exclusion Criteria:

* History of developmental delay or disorders
* History of any medical conditions ( that may impact the development)

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Local population; children and adolescents
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Perceptual organization index- Matrix reasoning subtest | 10-15 minutes
  The examinee views an incomplete matrix or series and selects the response option that completes the matrix or series. Scoring is based on whether the response is right or wrong.
Perceptual organization index- Block design subtest | 15-20 minutes
  The Block Design subtest is designed to measure the ability to analyze and synthesize abstract visual stimuli. While viewing a constructed model or a picture in the Stimulus Book, the examinee uses red- and-white blocks to re-create the design within a specified time limit. Scoring is based on how quickly the participant completes.
Processing speed index- Coding subtest | 2-3 minutes
  The processing speed index measures a child's ability efficiently to scan and understand visual information and complete a task with the data. Scoring is based on how many can the participant finish in 120 seconds.
Working memory index- Digit span subtest | 5-10 minutes
  The task digit span uses numbers. Memory span is a common measure of short-term memory. It is also a component of cognitive ability. Scoring is based on how many correct answers (recall) are achieved

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates